CLINICAL TRIAL: NCT01960062
Title: Impact of Web-based Care Management for Poorly Controlled Type 2 Diabetes Mellitus: a Randomized, Controlled Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no potential participants met the inclusion criteria
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GA-11NYate-01
Record Dates: First submitted 2013-09-24; First posted 2013-10-10 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; web-based; software; device
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Diabetes care with primary care practitioner supplemented with clinical pharmacy specialist
- Intervention (Experimental): Diabetes care with primary care practitioner and clinical pharmacy specialist, with the aid of a diabetes software and device to upload glucometer results from home
  Interventions: Device: Diabetes software and device

INTERVENTIONS:
Device: Diabetes software and device — USB cord, CD-rom, and application to allow communication with provider
  Arms: Intervention

SUMMARY:
Between October 1 and November 30, 2011, participants will be enrolled in this study comparing the use of MyLink web-based care with usual CPS care. Patients age 18- 74 with HbA1c ≥ 9% in the last 12 months will be identified. It is expected that approximately 32 people (16 per group) will participate in the study. Once eligible patients are found, they will be randomly assigned (like the flip of a coin) to usual care with the CPS or usual care with the CPS plus web-based care using the MyLink software. Participants using the software will agree to upload their glucometer measurements using the software every 2- 4 weeks. Following the receipt of the glucometer data, either electronically from intervention group participants or verbally from the control group participants, medications/ doses will be adjusted by the pharmacist as needed to achieve HbA1c goals. Participants in both groups will receive a follow-up HbA1c 2-4 months after enrollment to see if there were any significant changes in HbA1c between groups.

DETAILED DESCRIPTION:
Diabetes is an increasingly important public health issue. The American Diabetes Association estimates that 25.8 million people in the United States (8% of the total population) currently have diabetes. In fact, it is estimated that as many as 30.3 million Americans will have the disease by the year 2030. Concurrently, the economic impact of diabetes is rising at an alarming rate. In 2007, all costs associated with diabetes totaled $174 billion; $116 billion was spent on direct medical costs. Diabetes is associated with significant morbidity and mortality, a leading cause of blindness, kidney failure, stroke, and cardiovascular death.

Given the chronically progressive nature of diabetes, controlling the disease and preventing or delaying complications necessitates constant communication between the patient and the provider. Diabetes care limited to clinic visits does not meet the needs of many patients. With the increasing diabetes burden, there is an unmet need for innovative care methods. The internet's widespread availability has paved the way for increased utilization of web-based care management programs to manage chronic diseases such as diabetes mellitus.

A few randomized controlled trials have evaluated the use of web-based care in diabetes. These trials, ranging from 3 months to 30 months, have shown favorable changes in Hemoglobin A1c (HbA1c), as well as patient and provider satisfaction. A web-based application called MyLink has been used and evaluated in some Kaiser Permanente regions with impressive differences in HbA1c between groups utilizing web-based care versus usual care. This tool, along with appropriate software, enables patients to upload glucometer results from home, to the care provider in the office. Patients are able to view trends on their computer screen to see how lifestyle activities affect their blood sugar. The primary objective of this study is to evaluate the potential role of the MyLink web-based care management program in improving diabetes-related measures. It is expected that participants using web-based care will achieve a greater improvement in HbA1c than patients receiving usual care from the Clinical Pharmacy Specialist (CPS).

Between October 1 and November 30, 2011, participants will be enrolled in this study comparing the use of MyLink web-based care with usual CPS care. Patients age 18- 74 with HbA1c ≥ 9% in the last 12 months will be identified. It is expected that approximately 32 people (16 per group) will participate in the study. Once eligible patients are found, they will be randomly assigned (like the flip of a coin) to usual care with the CPS or usual care with the CPS plus web-based care using the MyLink software. Participants using the software will agree to upload their glucometer measurements using the software every 2- 4 weeks. Following the receipt of the glucometer data, either electronically from intervention group participants or verbally from the control group participants, medications/ doses will be adjusted by the pharmacist as needed to achieve HbA1c goals. Participants in both groups will receive a follow-up HbA1c 2-4 months after enrollment to see if there were any significant changes in HbA1c between groups.

ELIGIBILITY:
Inclusion Criteria:

* Receiving care from a PCP at the specified KPGA medical centers
* 18-74 years of age
* Type 2 Diabetes Mellitus (DM)
* Treated with insulin or willing to start insulin therapy
* Most recent HbA1c in the previous 12 months ≥ 9%
* Internet capability
* Actively enrolled or willing to enroll on www.kp.org
* English speaking

Exclusion Criteria:

* Having received care from an endocrinology specialty physician or Hospice/ Palliative Care within the last 3 months
* Enrolled in another research study
* Using an insulin pump
* Type 1 DM

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c | 2-4 months

SECONDARY OUTCOMES:
Hemoglobin A1c<9 | 2-4 months
Office visit time | 2-4 months
  time spent with participants during office visit

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Yates, PharmD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Georgia Region, Atlanta, Georgia, United States